CLINICAL TRIAL: NCT02769221
Title: Comparison of the Initial Intubation Success Rate Between Video Laryngoscope and Rigid Video Stylet in Patients Undergoing Cervical Spine Surgery
Brief Title: Intubation Success Rate_Rigid Video Stylet Vs Video Laryngoscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, MD, PhD, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rigid video stylet intubation
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optiscope (Experimental): Endotracheal intubation by rigid video stylet, manufactural named Optiscope.
  Interventions: Device: Rigid video stylet
- McGrath (Active Comparator): Endotracheal intubation by video laryngoscope, manufactural named McGrath.
  Interventions: Device: Video laryngoscope

INTERVENTIONS:
Device: Rigid video stylet
  Other Names: Optiscope
  Arms: Optiscope
Device: Video laryngoscope
  Other Names: McGrath
  Arms: McGrath

SUMMARY:
This study compare the intubation success rate between video laryngoscope and rigid video stylet in cervical spine surgery patients. Half of patients will receive endotracheal intubation by video laryngscope, other half of patients will receive endotracheal intubation by rigid video laryngoscope.

DETAILED DESCRIPTION:
Video laryngoscope and lightwand are widely used at endotracheal intubation in cervical spine patients.

Video laryngoscope is useful because of identification of anatomic structure around the oral cavity and vocal cord.

Rigid video stylet resemble lightwand, but it has a video at the end of stylet. So rigid video stylet is useful at confirmation of vocal cord.

ELIGIBILITY:
Inclusion Criteria:

* 20~80 years old adult patients, ASA class I-III
* Cervical spine surgery in general anesthesia

Exclusion Criteria:

* Patients who did not agree with the study
* History of GERD
* Congenital or acquired lesion like tumor, polyp, trauma, abcess, inflammation, foreign body
* Surgery of trachea or airway
* History of radiation around neck area
* Increased possibility of aspiration
* Coagulation abnormality

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of success rate between two groups | immediately

SECONDARY OUTCOMES:
Survey of blood tinged endotracheal tube, bleeding in oral cavity, hoarseness, sore throat | Within 24 hours after endotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Pyoung Park, MD, PhD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu CN, Ma WH, Wei JQ, Wei HF, Cen QY, Cai QX, Cao Y. Laryngoscope and a new tracheal tube assist lightwand intubation in difficult airways due to unstable cervical spine. PLoS One. 2015 Mar 24;10(3):e0120231. doi: 10.1371/journal.pone.0120231. eCollection 2015. PMID 25803435
- [Background] Aziz MF, Abrons RO, Cattano D, Bayman EO, Swanson DE, Hagberg CA, Todd MM, Brambrink AM. First-Attempt Intubation Success of Video Laryngoscopy in Patients with Anticipated Difficult Direct Laryngoscopy: A Multicenter Randomized Controlled Trial Comparing the C-MAC D-Blade Versus the GlideScope in a Mixed Provider and Diverse Patient Population. Anesth Analg. 2016 Mar;122(3):740-750. doi: 10.1213/ANE.0000000000001084. PMID 26579847
- [Background] Silverberg MJ, Li N, Acquah SO, Kory PD. Comparison of video laryngoscopy versus direct laryngoscopy during urgent endotracheal intubation: a randomized controlled trial. Crit Care Med. 2015 Mar;43(3):636-41. doi: 10.1097/CCM.0000000000000751. PMID 25479112
- [Background] Dong Y, Li G, Wu W, Su R, Shao Y. Lightwand-guided nasotracheal intubation in oromaxillofacial surgery patients with anticipated difficult airways: a comparison with blind nasal intubation. Int J Oral Maxillofac Surg. 2013 Sep;42(9):1049-53. doi: 10.1016/j.ijom.2013.01.027. Epub 2013 May 25. PMID 23712007
- [Background] Kasuya Y, Takahashi E, Nagai M, Ozaki M. [Comparison of Tracheal Intubation Performance between Macintosh Direct Laryngoscope and McGRATH(R) MAC Video Laryngoscope among Anesthesia Trainees]. Masui. 2015 Dec;64(12):1291-6. Japanese. PMID 26790337
- [Background] Choi JW, Kim JA, Jung HJ, Kim WH. Tracheal Intubation with a McGrath(R) Series 5 Video Laryngoscope by Novice Personnel in a Cervical-immobilized Manikin. J Emerg Med. 2016 Jan;50(1):61-6. doi: 10.1016/j.jemermed.2015.06.079. Epub 2015 Oct 1. PMID 26432080
- [Background] Ong J, Lee CL, Lai HY, Lee Y, Chen TY, Shyr MH. A new video intubating device: trachway intubating stylet. Anaesthesia. 2009 Oct;64(10):1145. doi: 10.1111/j.1365-2044.2009.06092.x. No abstract available. PMID 19735417
- [Background] Yang M, Kim JA, Ahn HJ, Choi JW, Kim DK, Cho EA. Double-lumen tube tracheal intubation using a rigid video-stylet: a randomized controlled comparison with the Macintosh laryngoscope. Br J Anaesth. 2013 Dec;111(6):990-5. doi: 10.1093/bja/aet281. Epub 2013 Aug 23. PMID 23975566
- [Background] Kim JK, Kim JA, Kim CS, Ahn HJ, Yang MK, Choi SJ. Comparison of tracheal intubation with the Airway Scope or Clarus Video System in patients with cervical collars. Anaesthesia. 2011 Aug;66(8):694-8. doi: 10.1111/j.1365-2044.2011.06762.x. Epub 2011 May 13. PMID 21564045
- [Background] Turkstra TP, Craen RA, Pelz DM, Gelb AW. Cervical spine motion: a fluoroscopic comparison during intubation with lighted stylet, GlideScope, and Macintosh laryngoscope. Anesth Analg. 2005 Sep;101(3):910-915. doi: 10.1213/01.ane.0000166975.38649.27. PMID 16116013